CLINICAL TRIAL: NCT03260530
Title: Overall Functional Evaluation After Amputation of the Lower Limb; Locomotion, Energy Efficiency and Strategies to Adapt to the Prosthesis
Acronym: PROTEOR
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: CASILLAS PROTEOR 2016
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Lower Limb Amputation
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Locomotor evaluation — collection of parameters associated with walking and balance in patients with their usual prosthesis and then equipped with the new prosthesis
Other: Questionnaires — Houghton's scale, PPA-LCI, ABC, QEP, SF-12, SAT-PRO, ESAT

SUMMARY:
It appears necessary to confront the reality of the contribution of technological progress in the creation of prostheses with the specific features of lower limb amputees. These contributions must be clearly identified in their different functional dimensions. This justifies a quantitative approach to the locomotor abilities of these patients, with regard to bioenergy parameters (consumption of oxygen while walking) and motor biomechanical parameters (quantified analysis of movement), so as to measure the real impact of the proposed prosthesis technology, as a complement to classical qualitative approaches.

In this context, Dijon CHU, thanks to its Technological Investigation Platform (PIT, CIC 1432), and the company PROTEOR established a research partnership aiming to:

* Refine the indications for the prescription of new products, by ensuring that they correspond to the profiles of the patients concerned and their true needs,
* Study the underlying adaptive mechanisms, and establish new recommendations for their use, depending on the profiles of the users,
* And ultimately, better evaluate, in a more rigorous and systematic manner, the prostheses available on the market.

The research protocol presented in this document aims to provide a framework for part of the explorations that will be conducted in the context of this partnership. Lower-limb amputees who will be evaluated in this research will wear these prostheses (foot and/or knee prostheses), which bear the CE logo, and thus present all of the safety and performance conditions required for their use by these patients (prostheses destined for usual prescriptions), the objective of the study was not to evaluate the prostheses as such, but to explore and quantify the impact of these prostheses and their eventual modifications on the locomotor abilities of the patients concerned.

The investigations will be conducted using non-invasive evaluation tools available on the PIT platform, with no modification in the usual management of these voluntary patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to understand simple instructions, the fitting instructions and to provide informed consent
* Man or woman aged > 18 years)
* Lower-limb amputee, transtibial or transfemoral amputation

Exclusion Criteria:

* Adult under guardianship
* Subject without national insurance cover
* Pregnant or breast-feeding women
* Patients with hip desarticulation
* Subjects presenting severe associated diseases affecting gait

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients attending routine consultations for a prosthesis
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Evolution of self-selected gait speed test, before and after the change or modification of the prosthesis | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France